CLINICAL TRIAL: NCT07080502
Title: Construction and Evaluation of the Psychometric Properties of Vaginal Penetration Impairment Questionnaire
Brief Title: Vaginal Penetration Alteration Questionnaire
Acronym: CAPEVA
Status: Completed | Type: Observational
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Other Study IDs: cquezada01
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Female Sexual Dysfunction
Keywords: Assessment, Sexuality, Pain
MeSH Terms: conditions — Sexuality; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Application for the creation of a questionnaire on alterations in vaginal penetration — Development of domains and items:
  Through the judgment of 10 experts, the set of items of each domain will be identified.
  Development of the scale:
  A pilot will be carried out to guarantee the viability and feasibility of what was created in the previous stage; The questionnaire will be applied to 30. participants.
  Evaluation of the scale:
  At this stage, the Questionnaire will be applied to a larger sample: 10 participants for each item create. In the same way as the previous stage, the Female Sexual Function Index will be applied together with the created questionnaire.

SUMMARY:
Female sexual dysfunctions reach a prevalence of between 38 and 64%, where various factors are involved. One of the sexual dysfunctions that afflict women are those related to pelvic pain and penetration disorders that are closely related to feelings of anguish and anxiety.

Due to the absence of specific, validated and reliable evaluation tools, the purpose of this work is to create an evaluation instrument for women who suffer from this dysfunction, which is self-administered and where the health professional can obtain clear and precise information about his patient. For this, an observational, multicenter study will be carried out in the city of Toledo, Spain, which consists of three large stages; The first will be the creation of domains and items through expert judgment, then a pilot will be carried out to analyze the viability and feasibility and finally the three psychometric properties will be analyzed: validity, confidence and sensitivity to change.

DETAILED DESCRIPTION:
Questionnaires play an important role in practice and research, both as diagnostic clinical tools, measurement of treatment-induced changes, and as research tools when describing a study population and its sexual function. Having a specific, validated, reliable, self-reported tool could facilitate these areas and therefore improve the quality of life of women.

The main objective is:

To build a valid and reliable instrument that is easy to apply for the evaluation of alterations in vaginal penetration and genito-pelvic pain.

An observational, multicenter project is presented that consists of the construction and validation of a Questionnaire in Spanish on Results Perceived by Patients / Health-Related Patient Reported Outcomes.

In stage 1, 10 professionals will be invited to participate, constituting an expert judgment; In stage 2, the pilot will be carried out with 30 women and 2 professionals who can explain the questionnaire to the participants and who can answer questions; In stage 3, a sample size of 10 respondents per item prepared will be required.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 60 who present genito-pelvic pain and/or difficulty in sexual activities for a period of 3 months, incapacity and/or difficulty in penetrating some type of intravaginal device, presenting complaints or inability to intracavitary gynecological evaluation

Exclusion Criteria:

* Presence of urogynecological infections, vaginal postpartum less than 6 months and 3 months via cesarean section, pelvic surgeries less than 6 months old, cognitive alterations, having neurological problems, exclusive breastfeeding.

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: This project is aimed at women with complaints of discomfort during vaginal penetration, either during sexual activity, when placing an intravaginal device, or difficulty performing an intracavitary gynecological examination.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
✓ Build a valid and reliable instrument that is easy to apply for the evaluation of alterations in vaginal penetration and genito-pelvic pain. | 5 months
  To achieve this goal it is necessary to meet the 3 sub-goals mentioned below.

SECONDARY OUTCOMES:
Establish domains and items that will form the questionnaire for the evaluation of penetration disorders and genito-pelvic pain. | 30 days
  Through the judgment of 10 experts, the set of elements of each domain will be identified. These professionals will be physiotherapists, gynecologists, midwives and professionals who are experts in creating health scales or questionnaires. Twice as many items should be prepared as it is thought the questionnaire should have. It should be considered that the administration time of the questionnaire does not exceed 10 minutes. The response formats will be of 5 ordered categories where the patient will choose an alternative.
Evaluate the viability and feasibility in the samples of participants and professionals. | 45 days
  A pilot test will be carried out to guarantee the viability and feasibility of what was created in the previous stage, in addition to ensuring that the questions are significant and understandable; The questionnaire will be applied to a small pre-established sample of participants (n=30) and the answers given will be analyzed to determine the optimal number of items/domains. In the same interview, the Female Sexual Function Index will be applied and a document called "Feasibility of the questionnaire for patients" will be given to them with questions about clarity, comprehensibility and adaptation to their condition. In addition to this, other documents will be delivered to the professionals: one called "Feasibility of the questionnaire for professionals" will be provided to the professionals who supervise the administration of the questionnaires to assess the time it has taken the participants to complete the questionnaire or difficulties that have had.
Evaluate the valid and reliable of the created questionnaire | 60 days
  At this stage, the Questionnaire is applied to a larger sample: 10 participants for each item created.
  Statistical tests will be applied to analyze the psychometrics of this instrument. The big aspects to analyze at this stage are reliability, validity and responsiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Asunción Ferri Morales, PhD, Principal Investigator — University of Castilla-La Mancha
Locations (1):
- University of Castilla-La Mancha, Toledo, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No